CLINICAL TRIAL: NCT03107039
Title: Exploring the Effects of Strength Training on Depressive Symptoms and Cardiovascular Risk in Black Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 512156
Record Dates: First submitted 2017-03-22; First posted 2017-04-11 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): This arm will use a resistance exercise curriculum.
  Interventions: Behavioral: Exercise
- Health Education (Active Comparator): This arm will use health education curriculum.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Exercise — A 12 week resistance exercise curriculum
  Arms: Exercise
Behavioral: Health Education — A 12 week health education curriculum
  Arms: Health Education

SUMMARY:
This study will address a gap in the literature and advance the field of minority men's health. Specifically, it will be the first randomized controlled trial of resistance exercise as a dual intervention for depression symptoms and CVD risk reduction with depressed Black men.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing depression symptoms and generally healthy.

Exclusion Criteria:

* Anyone assessed to be unsafe to be enrolled.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Black or African American
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | 6 months
  The Quick Inventory of Depression Symptomatology will be used to assess depression.

SECONDARY OUTCOMES:
Blood lipids | 6 months
  Total cholesterol, HDL, LDL, and triglycerides will be assessed from a blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciccolo, PhD, Principal Investigator — Teachers College
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ciccolo JT, Louie ME, SantaBarbara NJ, Webster CT, Whitworth JW, Nosrat S, Chrastek M, Dunsiger SI, Carey MP, Busch AM. Resistance training for Black men with depressive symptoms: a pilot randomized controlled trial to assess acceptability, feasibility, and preliminary efficacy. BMC Psychiatry. 2022 Apr 21;22(1):283. doi: 10.1186/s12888-022-03935-x. PMID 35448974
- [Derived] Busch AM, Louie ME, SantaBarbara NJ, Ajayi AA, Gleason N, Dunsiger SI, Carey MP, Ciccolo JT. Effects of resistance training on depression and cardiovascular disease risk in Black men: Protocol for a randomized controlled trial. Ment Health Phys Act. 2019 Oct;17:100299. doi: 10.1016/j.mhpa.2019.100299. Epub 2019 Sep 12. PMID 32863882